CLINICAL TRIAL: NCT00517764
Title: The Role of Childhood Adversity and Genetic Polymorphisms in the Serotonin and Brain-Derived Neurotrophic Factor Systems in the Sensitization to Stress in First-Onset Major Depression (Blue Sky Project)
Brief Title: Childhood Adversity, Genetic Polymorphisms and Stress in First Onset Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Queen's University (Other)
Responsible Party: Principal Investigator, Kate Harkness, Research Scientist, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155/2006
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: major depressive disorder; MDD; escitalopram; open-label; major depression; serotonin transporter; brain-derived neurotrophic factor
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (No Intervention): Healthy matched control, no intervention
- Escitalopram (Active Comparator): Depressed subjects receiving escitalopram
  Interventions: Drug: escitalopram
- subjects with major depression (No Intervention): Depressed subjects not receiving study treatment, but taking part in study measures.

INTERVENTIONS:
Drug: escitalopram — Patients started on 20mg of escitalopram and this dose was increased based on tolerability and therapeutic response to a maximum dose of 40mg by week 12. The trial was 16 weeks. The treatment trial has completed and is no longer accepting patients.
  Other Names: Lexapro; Cipralex; S-citalopram
  Arms: Escitalopram

SUMMARY:
The Blue Sky Project, a 5-year study funded by the Canadian Institutes of Health Research, seeks to examine how genetics and early life experiences work together to cause a person's very first onset of depression by increasing sensitivity to stress.

DETAILED DESCRIPTION:
Many forms of stress can precipitate an episode of depression. However, not everyone who experiences these sorts of stressors becomes depressed. Individuals with an at-risk genetic profile are more likely to get depressed in the face of stress, and require less severe levels of stress to get depressed, than individuals without this genetic profile. This model can help explain why young people get depressed the very first time. Young people with a particular variant of the serotonin transporter gene might require less severe levels of stress in both childhood and adulthood to precipitate their first episode of depression than individuals who do not possess this at-risk genetic variant. The current study involves 3 arms:

Participants at the Centre for Addiction and Mental Health site were enrolled in a 16-week trial of escitalopram (Lexapro/Cipralex), an established SSRI antidepressant that has been shown to be more effective and tolerable than other SSRIs. A psychiatrist and a trained research assistant will meet with participants every 2-3 weeks for the duration of the 16-week trial and participants will be asked to complete a number of standard psychological tests. After completion of the treatment phase, participants may continue into the follow-up phase involving monthly telephone contact and short appointments over an 18-month period. This arm of the study has finished and is no longer recruiting participants.

Participant at the Sunnybrook Health Sciences Centre site were enrolled in an assessment-only non-treatment arm. A research assistant met with participants to complete the same standard psychological tests as above. Participants received standard medical care from their attending psychiatrist. Participants may continue into the follow-up phase involving short appointments over an 18-month period to complete psychological assessments. This arm of the study has finished and is no longer recruiting participants.

Participant at the Queen's University site are enrolled in an assessment-only non-treatment arm. A research assistant will meet with participants to complete the same standard psychological tests as above. Participants will receive standard medical care from their attending psychiatrist or will be referred for treatment if they do not currently have a psychiatrist. Participants may continue into the follow-up phase involving short appointments over an 18-month period to complete psychological assessments.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of non-psychotic unipolar major depression; first onset
* Between 16 and 29 years of age
* Free of antidepressant treatment for a minimum of two weeks prior to treatment OR on an inadequate antidepressant treatment
* Minimum 8th grade education and fluency in reading English
* Live in the Kingston Area; willing to travel to the Queen's University for appointments

Exclusion Criteria:

* Diagnosis of previous episode(s) of major depression
* Past or present diagnosis of Bipolar Disorder, Schizoaffective Disorder, Schizophrenia, Substance Dependence Disorder, Borderline Personality Disorder, Anti-social Personality Disorder, or Organic Brain Syndrome
* Electroconvulsive Therapy in the past 6 months
* Concurrent serious medical illness judged to be contributing to the depression or impacting on treatment
* Presence of significant suicidal ideation

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 299 (Actual)
Dates: Start 2006-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRDS) | every 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kate L Harkness, PhD, Principal Investigator — Queens University; R.Michael Bagby, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Queens University, Kingston, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research